CLINICAL TRIAL: NCT03952468
Title: Combined Transcranial Magnetic Stimulation and Brief Cognitive Therapy to Reduce Suicide Behavior in High-Risk Veterans
Brief Title: Combined TMS and Brief Cognitive Behavioral Therapy to Reduce Suicide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIR 17-201
Record Dates: First submitted 2019-05-03; First posted 2019-05-16 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Suicide
Keywords: suicide prevention; Veterans
MeSH Terms: conditions — Suicide; Suicide Prevention | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: 130 Veterans admitted to the Providence VAMC psychiatric inpatient unit due to suicide attempt or ideation with intent to make an attempt will be recruited and randomly assigned to receive: a) active TMS+BCBT or b) sham TMS+BCBT. Both interventions will begin within the week following hospital discharge, and Veterans will be followed for 12 months post-discharge.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Prior to each TMS session, un-blinded study staff will attach the appropriate (i.e., active or sham) coil according to the participants' randomization code (obtained from the urn randomization computer program). This will facilitate "triple blind" stimulation, where the participant, TMS provider, and outcome rater are blind to group assignation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TMS + Brief Cognitive Behavioral Therapy (Active Comparator): Combined transcranial magnetic stimulation and brief cognitive behavioral therapy for suicide
  Interventions: Device: Transcranial Magnetic Stimulation; Other: Brief Cognitive Behavioral Therapy
- Sham TMS + Brief cognitive behavioral therapy (Sham Comparator): Sham Transcranial magnetic stimulation and brief cognitive behavioral therapy for suicide
  Interventions: Device: Transcranial Magnetic Stimulation; Other: Brief Cognitive Behavioral Therapy

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Administration of rapidly fluctuating magnetic field, delivered over the dorsolateral prefrontal cortex.
  Other Names: TMS
Other: Brief Cognitive Behavioral Therapy — BCBT is a well-established and efficacious treatment that is an extension of Cognitive Behavioral Therapy, a treatment that is widely implemented across VA health care systems.

SUMMARY:
High rates of Veteran suicide remain a tragedy. Rates of Veteran suicide have not decreased for 10 years, despite the best efforts of the field. Those interventions that do exist have only modest effects, which are simply insufficient for the magnitude of the problem. This proposal will combine two treatments - brief cognitive behavioral therapy (BCBT) and repetitive transcranial magnetic stimulation (TMS). Both of these interventions can reduce suicide and are available at Veterans Affairs Medical Centers across the country, yet to date no one has combined these therapies. This proposal will test the effect of this combination, and, if successful, will lead to a novel yet implementable new treatment to reduce Veteran suicide.

DETAILED DESCRIPTION:
The goal of the proposed study is to test the effect of adding Transcranial Magnetic Stimulation (TMS) to Brief Cognitive Behavioral Therapy (BCBT) to reduce Veterans' rates of suicide ideation and related behaviors. Over 20 Veterans die each day of suicide and rates have not appreciably decreased in the last ten years.

BCBT is a well-established and efficacious treatment that is an extension of Cognitive Behavioral Therapy, a treatment that is widely implemented across VA health care systems. However, not all patients respond to BCBT. Thus finding ways to enhance treatment efficacy for reducing suicide is critical. Transcranial Magnetic Stimulation (TMS) may be an optimal treatment to use in conjunction with psychotherapy. TMS is a noninvasive technique that uses a pulsed magnetic field to induce neuronal depolarization in a targeted brain region, typically the left dorsolateral prefrontal cortex. TMS can reduce psychiatric symptoms associated with suicide risk in Veterans, including depression and PTSD. Furthermore, TMS is not associated with the systemic and costly side effects associated with medications used for these disorders (e.g., weight gain, diabetes, sexual side effects).

The primary objective of this study is to conduct a fully-powered randomized controlled trial evaluating the effect of adding a standard TMS course of treatment to BCBT to reduce suicide behaviors in a sample of Veterans hospitalized for suicide behavior. One hundred and thirty (130) Veterans admitted to the psychiatric unit for suicide ideation or attempts will be randomly assigned to either active TMS plus BCBT or to sham TMS plus BCBT. Participants will be assessed at baseline, post treatment, six, and 12 months post hospital discharge. Efficacy of the program will be determined by examining a primary suicide composite outcome and several secondary outcomes including suicide attempt, time to first attempt, number of re-hospitalizations and severity and severity of suicidal ideation. Secondary analyses will be conducted to help identify the types of patients who will receive the most benefit from the addition of TMS to BCBT Brief Cognitive Behavioral Therapy for suicide.

If successful, this study would result in a combined treatment to decrease suicide ideation and related behaviors. The proposal addresses HSRD post-deployment health priority, specifically suicide prevention and is innovative in that it will be the first study to examine efficacy of combined treatment specifically for suicide prevention.

ELIGIBILITY:
Inclusion Criteria:

-Suicide attempt or suicidal ideation with intent to make a suicide attempt within 48 hours of hospitalization as indicated on the hospital chart and confirmed by administration of the C-SSRS.

Exclusion Criteria:

* Primary psychotic disorder
* Bipolar disorder
* Cognitive impairment which would interfere with adequate participation in the project (MMSE < 20).
* For safety, participants must meet established screening criteria safety during MRI, which is implemented as a conservative measure given the application of TMS in this population, since MRI involves magnetic fields at similar intensity to those emitted from the stimulation coil. These measures require a patient not having the following (unless MRI-safe):

  * Cardiac pacemaker
  * Implanted device (deep brain stimulation) or metal in the brain, cervical spinal cord, or upper thoracic spinal cord.
* TMS-specific exclusions are:

  * pregnancy/lactation, or planning to become pregnant during the study
  * lifetime history of moderate or severe traumatic brain injury (TBI)
  * Current unstable medical conditions
  * Current (or past if appropriate) significant neurological disorder
  * Lifetime history seizure disorder
  * Primary or secondary CNS tumors
  * Stroke
  * Cerebral aneurysm.
  * Other exclusions are conditions that would like to be worsened by TMS, such as bipolar disorder
  * Place Veterans at greater risk of seizures from TMS, such as severe and uncontrolled substance use disorder
  * Inability to participate in CBT
  * Other conditions or circumstance that, in the opinion of the investigator team, has the potential to prevent study completion and/or to have a confounding effect on outcome assessments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Primack, PhD MA, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (1):
- Providence VA Medical Center, Providence, RI, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bozzay ML, Primack J, Barredo J, Philip NS. Transcranial magnetic stimulation to reduce suicidality - A review and naturalistic outcomes. J Psychiatr Res. 2020 Jun;125:106-112. doi: 10.1016/j.jpsychires.2020.03.016. Epub 2020 Mar 28. PMID 32251917
- [Result] Barredo J, Bozzay ML, Primack JM, Schatten HT, Armey MF, Carpenter LL, Philip NS. Translating Interventional Neuroscience to Suicide: It's About Time. Biol Psychiatry. 2021 Jun 1;89(11):1073-1083. doi: 10.1016/j.biopsych.2021.01.013. Epub 2021 Feb 1. PMID 33820628
- [Result] Bozzay ML, Jiang L, Zullo AR, Riester MR, Lafo JA, Kunicki ZJ, Rudolph JL, Madrigal C, Clements R, Erqou S, Wu WC, Correia S, Primack JM. Mortality in patients with heart failure and suicidal ideation discharged to skilled nursing facilities. J Geriatr Cardiol. 2022 Mar 28;19(3):198-208. doi: 10.11909/j.issn.1671-5411.2022.03.009. No abstract available. PMID 35464651
- [Derived] Bozzay ML, Primack JM, Swearingen HR, Barredo J, Philip NS. Combined transcranial magnetic stimulation and brief cognitive behavioral therapy for suicide: study protocol for a randomized controlled trial in veterans. Trials. 2020 Nov 12;21(1):924. doi: 10.1186/s13063-020-04870-6. PMID 33183345

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following enrollment, 22 Veterans were not randomized. Of these 22 Veterans, 7 were ineligible, 6 were lost to contact, and 9 requested to withdraw participation due to starting residential treatment or work/scheduling concerns.
Groups:
- Active TMS + Brief Cognitive Behavioral Therapy: Combined transcranial magnetic stimulation and brief cognitive behavioral therapy for suicide
  Transcranial Magnetic Stimulation: Administration of rapidly fluctuating magnetic field, delivered over the dorsolateral prefrontal cortex.
  Brief Cognitive Behavioral Therapy: BCBT is a well-established and efficacious treatment that is an extension of Cognitive Behavioral Therapy, a treatment that is widely implemented across VA health care systems.
Period: Overall Study
Arm/Group | Active TMS + Brief Cognitive Behavioral Therapy | Sham TMS + Brief Cognitive Behavioral Therapy
Started | 18 (One participant was randomized, but discontinued by PI prior to start of TMS treatment due to substance use.) | 15
Completed TMS+BCBT Phase | 15 (Two withdrew during the TMS+BCBT phase due to diminished availability in schedule. One completed TMS #8 and Therapy #1 and the other completed TMS #10 and Therapy #1.) | 12 (One withdrew during the TMS+BCBT phase due to diminished availability in schedule after completing TMS #28 and Therapy #5. One was lost to contact after completing TMS #10 and Therapy #2. One requested to stop TMS after #21 due to perceived lack of efficacy, but continued with therapy. This participant died by suicide after Therapy #5.)
Completed BCBT-Only and Endpoint Assessments | 14 (One completed 6 therapy sessions but was lost to contact.) | 12
Completed 6-month Follow-up | 12 (Two were lost to contact and did not complete 6-month follow-up.) | 11 (One was lost to contact and did not complete 6-month follow-up.)
Completed 12-month Follow-up | 12 | 8 (Three did not complete 12-month follow-up. Of these, two were lost to contact and one was re-hospitalized with suicidal ideation with a plan the day the follow-up was scheduled.)
Completed | 12 | 8
Not Completed | 6 | 7
Not completed — Death | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 3 | 4
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active TMS + Brief Cognitive Behavioral Therapy | Sham TMS + Brief Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 18 | 15 | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] — Demographics self-report. Text box
  Years | 47.8 (10.9) | 50.4 (13.6) | 49.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 15 | 13 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 15 | 32
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 15 | 12 | 27
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 15 | 33
CSSRS ideation severity, past two weeks [Mean (Standard Deviation); unit: units on a scale (0-5)] — Columbia Suicide Severity Rating Scale, ideation subscale for past two weeks. Scores range from 0-5 with higher scores representing more severe ideation.
  units on a scale (0-5) | 4.56 (0.51) | 4.33 (0.62) | 4.45 (0.56)
CSSRS past two week attempts [Mean (Standard Deviation); unit: number of attempts] — Past two weeks number of reported suicide attempts collected via interview using the CSSRS suicide attempt item.
  number of attempts | 0.39 (0.70) | 0.27 (0.80) | 0.33 (0.74)
CSSRS past two week behavior composite [Mean (Standard Deviation); unit: number of suicide behaviors] — Past two week report on CSSRS interview. Count of number of suicide attempts, aborted attempts, and interrupted attempts.
  number of suicide behaviors | 0.61 (0.92) | 0.33 (0.82) | 0.48 (0.87)
CSSRS ideation severity, lifetime [Mean (Standard Deviation); unit: units of a scale] — Columbia Suicide Severity rating scale - Ideation subscale interview for lifetime most severe ideation on a scale of 0-5 with higher scores representing more severe ideation type.
  units of a scale | 4.56 (0.51) | 4.4 (0.51) | 4.48 (0.51)
CSSRS (Lifetime number of attempts) [Mean (Standard Deviation); unit: number of attempts] | 2.78 (5.93) | 5.47 (8.33) | 4.00 (7.13)
CSSRS lifetime total number of suicide behaviors composite [Mean (Standard Deviation); unit: number of behaviors] — Total lifetime number of interrupted, aborted, and actual attempts reported on the CSSRS interview.
  number of behaviors | 2.94 (5.89) | 6.53 (9.98) | 4.58 (8.08)
Beck Hopelessness Scale (BHS) [Mean (Standard Deviation); unit: units on a scale] — THE BHS is a 20-item self-report measure designed to measure three major aspects of hopelessness: feelings about the future, loss of motivation, and expectation. Items are rated as true/false with true responses scored as 1 point. Scoring ranges from 0-20 with the following scale 0-3: normal, 4-8: mild hopelessness, 9-14: moderate hopelessness, and 15-20: severe hopelessness. Total scores were used for this study with higher scores indicative of greater hopelessness.
  units on a scale | 11.5 (6.71) | 11.0 (6.46) | 11.27 (6.50)
Brief Symptom Inventory (BSI): Psychiatric Symptoms [Mean (Standard Deviation); unit: Mean score (GSI)] — The BSI is a 53-item self-report questionnaire developed by Derogatis and Melisarotos to measure psychological distress and assess the severity of symptom across the following dimensions: Somatization, Obsession-compulsion, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism. Items are rated on a 5-point Likert scale from 0-4. The Global severity index (GSI) was used and reported. GSI is a mean score for all items across all dimensions. Higher scores are indicative of greater psychological distress.
  Mean score (GSI) | 2.10 (1.13) | 1.85 (1.04) | 1.99 (1.08)
PTSD Checklist [Mean (Standard Deviation); unit: units on a scale] — The PCL-5 is a 20-item self report measure that assesses the DSM-5 symptoms of PTSD on a 5-point Likert scale (0-4). Total symptom severity score is obtained by summing the scores for all 20 items (0-80). Higher scores are indicative of greater severity.
  units on a scale | 49.11 (20.46) | 43.67 (23.79) | 46.64 (21.86)
Inventory of Depressive Symptomatology-Self Report (IDS-SR) [Mean (Standard Deviation); unit: units on a scale] — The IDS-SR is a 30-item self report measure designed to assess the severity of depressive symptom over the last week. Items are scored using a 4-point Likert scale ranging from 0-3 with higher scores indicating greater severity. Total scores are calculated by summing responses to 28 items to obtain a total score ranging from 0-84.
  units on a scale | 44.0 (17.44) | 39.87 (15.71) | 42.12 (26.80)
AUDIT-10 (Alcohol Use Disorders Identification Test) [Mean (Standard Deviation); unit: units on a scale] — The AUDIT is a 10-item screening tool developed by the World Health organization to assess alcohol consumption, behaviors, and problems associated with alcohol use. Individual items are rated on a 5-point Likert scale ranging from 0-4 with higher scores indicating more severe use. Range of possible scores is 0-40 with higher scores indicating more severe alcohol use/behaviors.
  units on a scale | 9.83 (11.98) | 9.47 (11.58) | 9.67 (11.62)
DUDIT (Drug Use Disorders Identification Test) [Mean (Standard Deviation); unit: units on a scale] — the DUDIT is an 11-item self report measure used to assess drug use and behaviors. Items 1-9 are scored on a 0-4 Likert scale and items 10-11 are scored 0, 2, 4. Total scores are the summation of all items and range from 0-44 with higher scores indicating greater severity of drug-use-related problems.
  units on a scale | 4.67 (6.51) | 2.80 (4.00) | 3.82 (5.51)
World Health Organization Disability Assessment Schedule (WHODAS-2.0) [Mean (Standard Deviation); unit: standardized scores] — The WHO-DAS 2.0 36-self-version is a 36-item measure that assesses disability across six domains of functioning (cognition, mobility, self-care, getting along, life activities, and participation) in adults. Each item is rated on a 5-point likert scale from 0-4 with higher scores indicating greater disability. Total score is calculated by summing the item scores and then converted into a standardized score ranging from 0-100 with higher scores indicating greater disability.
  standardized scores | 50.89 (30.20) | 48.20 (23.03) | 49.67 (26.20)
Beck Scale for suicide ideation (BSSI) [Mean (Standard Deviation); unit: units on a scale] — The BSSI is a 19-item measure designed to assess the severity of suicidal thoughts in the week prior to evaluation. Each item is scored based on an ordinal scale from 0-2 and the total score range is 0-38 with higher scores indicating greater severity.
  units on a scale | 15.83 (8.45) | 16.13 (4.42) | 15.97 (6.82)
McLean Borderline Personality screen (MSI-BPD) [Count of Participants; unit: Participants] — The MSI-BPD is a 10-item self-report tool designed to screen for Borderline Personality. Each item is rating on a dichotomous scale (1 for present, 0 for absent) and the total score ranges from 9-10 with higher scores indicative of greater likelihood for the presence of BPD. In this study, count is reported for the number of participants who scored >= 7 (the cutoff indicating presence of BPD symptoms).
  Participants | 13 | 8 | 21
SCID Module A [Count of Participants; unit: Participants]
  Current Major Depressive Episode | 14 | 13 | 27
  Past Major Depressive Episode | 2 | 1 | 3
  Current Hypomanic Episode | 0 | 0 | 0
  Past Hypomanic Episode | 0 | 0 | 0
  Did not meet diagnostic criteria | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Columbia Suicide Severity Rating Scale (CSSRS) (Suicide Composite)
Description: The Columbia suicide severity rating scale is an interview-administered assessment of suicide ideation and behavior. The full CSSRS interview consists of two subscales, an ideation and behavior subscale. The primary outcome measure for this study utilized the behavior subscale.
  A study-created composite score was calculated by adding the total number of: 1) suicide attempts, 2) interrupted attempts, and 3) aborted attempts in the specified time frame. At baseline total number of behaviors covered lifetime number of total behaviors prior to baseline. Each subsequent assessment period assesses total number of behaviors since time of last assessment (e.g., endpoint = total number of behaviors from baseline to end of 12-week BCBT course, 6-month follow up = total number of behaviors from endpoint to 6 months post-baseline, 12 months = total number of behaviors from 6 month follow up to 12 month follow up.
Time Frame: Baseline, endpoint (end of 12-week BCBT course), 6-month follow-up, and 12 month follow up
Population: Due to study attrition, the number of participants at follow-up differs from the number of participants at baseline. See participant flow for more details.
Measure: Mean (Standard Deviation); unit: total number of suicide behaviors
Arm/Group | TMS + Brief Cognitive Behavioral Therapy | Sham TMS + Brief Cognitive Behavioral Therapy
Number analyzed (Participants) | 18 | 15
total number of suicide behaviors
  Baseline | 0.61 (0.92) | 0.33 (0.82)
  Endpoint (~12-weeks): number analyzed (Participants) | 14 | 12
  Endpoint (~12-weeks) | 0 (0) | 0.17 (0.39)
  6-Month Follow-Up: number analyzed (Participants) | 12 | 11
  6-Month Follow-Up | 0.08 (0.29) | 0.18 (0.40)
  12-Month Follow-Up: number analyzed (Participants) | 12 | 8
  12-Month Follow-Up | 0 (0) | 0 (0)

2. Secondary Outcome: Beck Scale for Suicide Ideation (BSSI)
Description: The BSSI is a 21-item measure designed to assess the severity of suicidal thoughts in the week prior to evaluation. The first 5 items are screeners (wish to live, wish to die, and desire to attempt suicide), followed by 14 items to assess suicidal risk factors. The last 2 items capture previous suicide attempts.
  Each item is scored based on an ordinal scale from 0-2 and the total score range is 0-38 with higher scores indicating greater severity.
  The SSI total score is obtained by adding up the ratings (0-2) from the first 19 items.
Time Frame: Baseline, endpoint (end of 12-week BCBT course), 6-month follow-up, and 12 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active TMS + Brief Cognitive Behavioral Therapy | Sham TMS + Brief Cognitive Behavioral Therapy
Number analyzed (Participants) | 18 | 15
units on a scale
  Baseline | 15.83 (8.45) | 16.13 (4.42)
  Endpoint (~12 weeks): number analyzed (Participants) | 14 | 12
  Endpoint (~12 weeks) | 5.14 (6.71) | 7.00 (5.24)
  6-Month Follow-Up: number analyzed (Participants) | 12 | 11
  6-Month Follow-Up | 5.17 (7.88) | 5.82 (8.81)
  12-Month Follow-Up: number analyzed (Participants) | 12 | 8
  12-Month Follow-Up | 4.33 (4.92) | 6.87 (6.10)

3. Secondary Outcome: The Longitudinal Interval Follow-up Evaluation (LIFE): Psychiatric Status Rating Scale for Suicidal Ideation
Description: The Longitudinal Interval Follow-up Evaluation (LIFE) is a timeline follow up interview measure that is administered at each of the assessment period. Participants are asked to describe their weekly suicidal thoughts and interviewers rate them on a 6-point Likert score ranging from 1 (not at all) to 6 (Extreme: has made preparations for a potentially serious suicide attempt). Data is then converted into the presence/absence of suicidal thoughts for each week of the follow up period. Data reported includes the mean number of weeks with reported suicidal thoughts (scores above 2).
Time Frame: Endpoint (end of 12-week BCBT course), 6-month follow-up, and 12 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of weeks with suicidal ideation
Arm/Group | Active TMS + Brief Cognitive Behavioral Therapy | Sham TMS + Brief Cognitive Behavioral Therapy
Number analyzed (Participants) | 14 | 12
number of weeks with suicidal ideation
  Endpoint | 9.21 (5.92) | 11.58 (7.01)
  6-Month Follow-Up: number analyzed (Participants) | 12 | 11
  6-Month Follow-Up | 5.92 (6.23) | 7.73 (7.48)
  12-Month Follow-Up: number analyzed (Participants) | 12 | 8
  12-Month Follow-Up | 11.00 (11.11) | 13.13 (12.00)

4. Secondary Outcome: Change in World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0)
Description: The WHODAS 2.0 is a 36-question, self-administered questionnaire and generic assessment instrument for health and disability that covers six domains: Cognition (items 3 and 6), Mobility (items 1 and 7), Self-care (items 8 and 9), Getting Along (items 10 and 11), Life Activities (items 2 and 12), and Participation (items 4 and 5). Items are rated from "None," "Mild," "Moderate," "Severe," to "Extreme or cannot do," indicating difficulty over the past month. Total score is calculated by summing the item scores and then converted into a standardized score ranging from 0-100 with higher scores indicating greater disability.
Time Frame: Baseline, endpoint (end of 12-week BCBT course), 6-month follow-up, and 12 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS + Brief Cognitive Behavioral Therapy | Sham TMS + Brief Cognitive Behavioral Therapy
Number analyzed (Participants) | 18 | 15
score on a scale
  Baseline | 50.89 (30.20) | 48.20 (23.03)
  Endpoint: number analyzed (Participants) | 14 | 12
  Endpoint | 35.36 (24.58) | 47.75 (22.63)
  6-Month Follow-Up: number analyzed (Participants) | 12 | 11
  6-Month Follow-Up | 34.92 (25.69) | 37.82 (21.03)
  12-Month Follow-Up: number analyzed (Participants) | 12 | 8
  12-Month Follow-Up | 34.83 (26.37) | 40.50 (31.87)

5. Secondary Outcome: Treatment History Interview THI: Emergency Services
Description: The THI is an interview used to collect information about psychotherapy, hospitalizations, medical treatment, pharmacotherapy, and other means of psychologically-related help that a person may use. For this study we assessed the use of emergency services (emergency room visits for psychiatric reasons and hospitalizations for psychiatric reasons). Outcome was the number of times a participant used either emergency department or was hospitalized for mental health reasons.
Time Frame: Endpoint (following a 12-week course of BCBT), 6-month follow-up, 12-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of times used emergency services
Arm/Group | Active TMS + Brief Cognitive Behavioral Therapy | Sham TMS + Brief Cognitive Behavioral Therapy
Number analyzed (Participants) | 14 | 12
number of times used emergency services
  Endpoint (12-weeks) | 0.14 (0.53) | 0.00 (0.00)
  6-Month Follow-Up: number analyzed (Participants) | 12 | 11
  6-Month Follow-Up | 0.08 (0.29) | 0.18 (0.60)
  12-Month Follow-Up: number analyzed (Participants) | 12 | 8
  12-Month Follow-Up | 0.42 (0.67) | 0.13 (0.35)

6. Secondary Outcome: Brief Symptom Inventory: Psychiatric Symptoms
Description: The BSI is a 53-item self-report questionnaire developed by Derogatis and Melisarotos to measure psychological distress and assess the severity of symptom across the following dimensions: Somatization, Obsession-compulsion, interpersonal sensitivity , depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism. Items are rated on a 5-point Likert scale from 0-4. The Global severity index (GSI) was used and reported. GSI is a mean score for all items across all dimensions. Higher scores are indicative of greater psychological distress.
Time Frame: Baseline, endpoint (end of 12-week BCBT course), 6-month follow-up, and 12 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Mean score (GSI)
Arm/Group | Active TMS + Brief Cognitive Behavioral Therapy | Sham TMS + Brief Cognitive Behavioral Therapy
Number analyzed (Participants) | 18 | 15
Mean score (GSI)
  Baseline | 2.10 (1.13) | 1.85 (1.04)
  Endpoint (12-weeks): number analyzed (Participants) | 14 | 12
  Endpoint (12-weeks) | 1.10 (0.87) | 1.47 (1.07)
  6-Month Follow-Up: number analyzed (Participants) | 12 | 11
  6-Month Follow-Up | 1.30 (0.99) | 1.27 (0.99)
  12-Month Follow-Up: number analyzed (Participants) | 12 | 8
  12-Month Follow-Up | 1.06 (0.79) | 1.18 (0.98)

ADVERSE EVENTS:
Time Frame: Up to one year.
Description: Adverse events as defined in our study were identical to clinicaltrials.gov definitions.
  Adverse events were collected in several ways: 1) events spontaneously reported by participants, 2) review of medical records preceding each follow up period, 3) systematically assessed through a side effects questionnaire that was administered before and after each TMS or sham TMS session, and 4) systematically assessed through the Treatment History Questionnaire.
Groups:
- Sham TMS + Brief Cognitive Behavioral Therapy: Sham Transcranial magnetic stimulation and brief cognitive behavioral therapy for suicide
  Sham Transcranial Magnetic Stimulation
  Brief Cognitive Behavioral Therapy: BCBT is a well-established and efficacious treatment that is an extension of Cognitive Behavioral Therapy, a treatment that is widely implemented across VA health care systems.
Arm/Group | TMS + Brief Cognitive Behavioral Therapy | Sham TMS + Brief Cognitive Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/18 | 1/15
Serious Adverse Events (participants affected / at risk) | 6/18 | 5/15
Other Adverse Events (participants affected / at risk) | 11/18 | 6/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMS + Brief Cognitive Behavioral Therapy (N=18) | Sham TMS + Brief Cognitive Behavioral Therapy (N=15)
Psychiatric rehospitalization (Psychiatric disorders) | 3 (4) | 2 (3) — Psychiatric rehospitalization due to suicide ideation or behaviors
Medical hospitalization (Surgical and medical procedures) | 1 (1) | 0 (0) — Hospitalization due to surgery or other medical procedures
Psychiatric hospitalization due to worsening mental health symptoms (Psychiatric disorders) | 1 (1) | 0 (0) — Psychiatric admission due to mental health symptoms (not SI/SB)
Medical hospitalization (Vascular disorders) | 0 (0) | 1 (1)
Medical hospitalization (General disorders) | 0 (0) | 2 (2)
ER visit for psychiatric reasons (Psychiatric disorders) | 1 (1) | 0 (0) — Visit to ER for psychiatric symptoms other than SI/SB
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMS + Brief Cognitive Behavioral Therapy (N=18) | Sham TMS + Brief Cognitive Behavioral Therapy (N=15)
Headaches (General disorders) | 3 (3) | 3 (3)
Treatment site discomfort (General disorders) | 10 (10) | 3 (3)

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic significantly impacted recruitment and retention particularly as inpatient psychiatric units shifted to house chronically ill patients and discharge planning moved to non-local environments. The requirement for daily stimulation visits for 6-8 weeks also impacted outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT03952468/Prot_SAP_001.pdf
  • Informed Consent Form (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT03952468/ICF_000.pdf